CLINICAL TRIAL: NCT02081131
Title: A Prospective Randomized Controlled Trial Comparing Laparoscopic Versus Open Pancreatoduodenectomy for Malignant Periampullary and Pancreatic Head Lesions
Brief Title: Pancreatic Head and Peri-ampullary Cancer Laparoscopic vs Open Surgical Treatment Trial (PLOT)
Acronym: PLOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLOT; CTRI/2013/09/004016 (Registry Identifier: Clinical Trials Registry India)
Record Dates: First submitted 2014-01-30; First posted 2014-03-07 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Adenocarcinoma of Head of Pancreas; Cholangio Carcinoma; Duodenal Adenocarcinoma; Carcinoma of Ampulla of Vater
Keywords: periampullary cancer; pancreatic cancer; randomized controlled trial; Whipple's operation; laparoscopy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Conversion to Open Surgery; Pancreaticoduodenectomy; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Surgery (Active Comparator): patients will be randomized to laparoscopic pancreatoduodenectomy group
  Interventions: Procedure: Laparoscopic surgery
- Open Surgery (Active Comparator): Patients will be randomized to Open pancreatoduodenectomy
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: Open surgery — pancreatic head resection by open method
  Other Names: Whipple's operation, pancreatoduodenectomy
  Arms: Open Surgery
Procedure: Laparoscopic surgery — laparoscopic pancreatoduodenectomy
  Other Names: laparoscopic pancreatoduodenectomy; whipple's operation; pylorus preserving pancreatoduodenectomy
  Arms: Laparoscopic Surgery

SUMMARY:
The aim of this study is to compare the two surgical approaches namely laparoscopic pancreatoduodenectomy and open pancreatoduodenectomy for management of periampullary and pancreatic head cancers in terms of parameters like hospital stay, pathological radicality, complication rate, peri-operative and post operative outcomes.

DETAILED DESCRIPTION:
Laparoscopic pancreatoduodenectomy (LPD) although technically difficult, requiring high degree of expertise, has shown equal efficacy in terms of complications, oncological safety & overall outcome to that of open pancreatoduodenectomy (OPD) with advantages of minimally invasive surgery like decreased blood loss, reduced pain, shorter hospital stay & early return to work.

Although current literature from various centres supports its use, the studies done so far are, case comparisons of either small sample of population or non-randomized trials. According to our knowledge, a randomized trial analyzing open versus laparoscopic pancreatoduodenectomy (PD) in terms of complications and outcome, has not been reported. With this current study we will try to address this issue.

This study is a prospective, randomized, parallel group, controlled trail comparing laparoscopic versus open pancreatoduodenectomy in relation to the hospital stay, peri-operative parameters, pathological radicality & complications.

This is a single institute based trial, being conducted at GEM hospital and research center, Coimbatore, TN, India. The trial has been approved by the GEM Hospital ethical committee.

Through this trial we are planning to enroll patients having resectable periampullary and pancreatic head malignant lesion at diagnosis. After full assessment, optimization, approval of hospital tumor board with informed consent, those patients selected for surgical therapy with curative intention, will be randomized using computer generated random numbers either into Laparoscopic Pancreatoduodenectomy (LPD) group or Open Pancreatoduodenectomy (OPD) group.

The details of surgery, blood loss, operating time, conversion if any as well as details of postoperative events, hospital stay & complications if any will be recorded in proforma. Protocols for adjuvant therapy according to pathological stages will be followed. These patients will be reviewed at 1, 3 and 6 months post-surgery.

The primary outcome will be hospital stay at time of discharge or death. The secondary outcomes will be Blood Loss, Operating Time, Complications and pathological radicality at discharge or death. The trial is expected to last for a duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females with a diagnosis of either of resectable Periampullary and pancreatic head cancers with

  1. No evidence of metastasis
  2. Radiological non-involvement of Superior Mesenteric Vein & Portal Vein
  3. Preserved fat planes between celiac axis, Hepatic Artery & Superior Mesenteric Artery

Exclusion Criteria:

1. Unresectable Tumor at surgery
2. Pancreatoduodenectomy for other diagnosis like cystic tumors or chronic calcific pancreatitis with head mass
3. With prior Neoadjuvant treatment

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hospital Stay | discharge from hospital or death which ever earlier recorded over 100 days from date of admission

SECONDARY OUTCOMES:
Blood loss | within 24 hours of primary surgical procedure
  Blood loss at surgery
Pathological radicality | within 7 days of surgery
  Two specimen arms will be compared on the basis of extent of pathological clearance like margin positivity rate, number of lymph nodes, average length of surgical margin
Operating time | At completion of the primary surgical procedure, recorded over 48 hrs
  Time calculated in minutes
Complication rate | 100 days from date of surgery
  Pancreatic surgery specific complications will be accessed by International Study group for pancreatic surgery ( ISGPS) classification like post operative pancreatic fistula ( POPF). Other complications will be accessed by Clavien Dindo Classification system

CONTACTS AND LOCATIONS:
Overall Officials: Senthilnathan Palanisamy, MS, DNB, Principal Investigator — Gem Hospital & Research Centre Private Limited, Coimbatore, Tamil Nadu, India; Palanivelu Chinnusamy, MS, MCh, Study Director — Gem Hospital & Research Centre Private Limited, Coimbatore, Tamil Nadu, India; Sandeep Sabnis, MS, Study Director — Gem Hospital & Research Centre Private Limited, Coimbatore, Tamil Nadu, India
Locations (1):
- Gem Hospital & Research Centre Private Limited, Coimbatore, Tamil Nadu, India

REFERENCES:
- [Background] Asbun HJ, Stauffer JA. Laparoscopic vs open pancreaticoduodenectomy: overall outcomes and severity of complications using the Accordion Severity Grading System. J Am Coll Surg. 2012 Dec;215(6):810-9. doi: 10.1016/j.jamcollsurg.2012.08.006. Epub 2012 Sep 19. PMID 22999327
- [Background] Palanivelu C, Rajan PS, Rangarajan M, Vaithiswaran V, Senthilnathan P, Parthasarathi R, Praveen Raj P. Evolution in techniques of laparoscopic pancreaticoduodenectomy: a decade long experience from a tertiary center. J Hepatobiliary Pancreat Surg. 2009;16(6):731-40. doi: 10.1007/s00534-009-0157-8. Epub 2009 Aug 4. PMID 19652900
- [Background] Kim SC, Song KB, Jung YS, Kim YH, Park DH, Lee SS, Seo DW, Lee SK, Kim MH, Park KM, Lee YJ. Short-term clinical outcomes for 100 consecutive cases of laparoscopic pylorus-preserving pancreatoduodenectomy: improvement with surgical experience. Surg Endosc. 2013 Jan;27(1):95-103. doi: 10.1007/s00464-012-2427-9. Epub 2012 Jun 30. PMID 22752284
- [Derived] Palanivelu C, Senthilnathan P, Sabnis SC, Babu NS, Srivatsan Gurumurthy S, Anand Vijai N, Nalankilli VP, Praveen Raj P, Parthasarathy R, Rajapandian S. Randomized clinical trial of laparoscopic versus open pancreatoduodenectomy for periampullary tumours. Br J Surg. 2017 Oct;104(11):1443-1450. doi: 10.1002/bjs.10662. PMID 28895142